CLINICAL TRIAL: NCT07092358
Title: Hereditary Ataxia Research on Multi-Omics and Neuroclinical Insights in the Yangtze Delta
Acronym: HARMONY
Status: Recruiting | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Collaborators: Huashan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-048-HARMONY
Record Dates: First submitted 2025-07-13; First posted 2025-07-29 (Actual); Last update posted 2025-07-29 (Actual); Status verified 2025-06

CONDITIONS: Hereditary Ataxia
Keywords: multiomics; clinical and genetic characteristics
MeSH Terms: conditions — Spinocerebellar Degenerations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — DNA, whole blood, serum, plasma, cerebrospinal fluid, saliva, skin fibroblasts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- HA Cohort: Patients with clinical suspected or genetic-confirmed hereditary ataxia
  Interventions: Other: None of intervention

INTERVENTIONS:
Other: None of intervention — No specific intervention was implemented in this study.

SUMMARY:
The goal of this observational study is to explore the clinical and genetic characteristics, multi-omics profiles, disease mechanisms, biomarkers, and potential therapeutic targets of hereditary ataxia (HA) in patients diagnosed with HA, primarily in the Yangtze River Delta region of China. The main questions it aims to answer are:

* What are the key pathogenic genetic variants, modifying factors and special inheritance patterns underlying HA?
* How do multi-omics profiles correlate with clinical phenotypes, disease progress and mechanism in HA patients?
* What are the implications of these findings for clinical practice?

Participants will:

* Undergo retrospective and prospective clinical data collection through long-term follow-up to observe disease onset, progression, and outcomes.
* Provide biological samples (e.g., blood, skin) to establish a biobank for multi-omics analyses.
* Be characterized using multidimensional omics technologies to identify disease-related molecular signatures, progression mechanisms, and potential regulatory targets.

DETAILED DESCRIPTION:
This project aims to establish a representative and continuously expanding cohort of hereditary ataxia in the Yangtze River Delta region of China. By integrating both retrospective and prospective study designs, the investigators will implement a observational ambispective cohort approach to comprehensively capture the natural history of the disease - including its onset, progression, and clinical outcomes - through systematic data collection from historical records and long-term follow-up of enrolled cases. In parallel, a biobank will be established by collecting biospecimens such as blood and skin samples from participants, providing high-quality biological materials for future research. Utilizing multi-omics technologies, including genomics, transcriptomics, epigenomics, etc., the investigators will explore key pathogenic genetic variants, disease-modifying factors, mechanisms underlying disease progression, biomarkers, and potential therapeutic targets. Through this integrated approach, the project is expected to significantly advance basic and translational research on hereditary ataxia, ultimately contributing to the development of precision diagnosis and effective intervention strategies for these debilitating neurodegenerative disorders.

ELIGIBILITY:
Inclusion Criteria:

* Presence of progressive ataxia as a primary or persistent clinical feature;
* Sufficient evidence to exclude acquired causes of ataxia (e.g., chronic intoxication, immune-mediated inflammation, acquired vitamin deficiency, acute injury, stroke, infection, or space-occupying disorders);
* For sporadic late-onset cases (≥30 years), disease duration must exceed 3 years, with no prominent progressive autonomic dysfunction or other features indicative of multiple system atrophy-cerebellar type (MSA-C);
* Ability and willingness of the participant or legal guardian to provide informed consent and complete the entire study process.

Exclusion Criteria:

* Patients whose causative genes identified through genetic testing and analysis do not fall within the defined spectrum of hereditary ataxias, based on consensus classifications from the MDS Task Force on Genetic Movement Disorders and the SRCA Working Group, along with current research advancements;
* Presence of concurrent cerebrovascular disease, brain tumors, or severe systemic illness;
* Refusal to sign informed consent or provide biological samples by the participant or legal representative;
* Inability or unwillingness to participate in follow-up assessments.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Chinese patients concentrated in the Yangtze River Delta region.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2035-06-30 (Estimated); Study Completion 2035-12-31 (Estimated)

PRIMARY OUTCOMES:
SARA scores | 10 years
  Scale for the Assessment and Rating of Ataxia (SARA) is a widely used tool specifically developed to quantify the severity of ataxia. It assesses multiple domains of ataxia, including gait, stance, sitting, speech, finger chase, nose-finger test, fast alternating hand movements, and heel-shin slide. It is applicable to patients with various forms of ataxia and provides a standardized method for tracking disease progression.
  * Minimum value: 0
  * Maximum value: 40
  * Interpretation: Higher scores indicate more severe ataxia (worse outcome).
ICARS scores | 10 years
  As a comprehensive assessment tool, International Cooperative Ataxia Rating Scale (ICARS) evaluates four main components of ataxia: postural and gait disturbances, limb ataxia, dysarthria, and oculomotor disorders. It is commonly used in clinical research and practice to measure the overall severity of ataxia, allowing for comparisons across different studies and patient populations.
  * Minimum value: 0
  * Maximum value: 100
  * Interpretation: Higher scores indicate more severe ataxia (worse outcome).
SDFS scores | 10 years
  Spinocerebellar Degeneration Functional Score (SDFS) focuses on assessing the functional status of patients with spinocerebellar degeneration by evaluating their ability to perform daily activities related to mobility. It ranges from 0 to 7：
  * 0: no functional handicap;
  * 1: no functional handicap but signs at examination;
  * 2: mild, able to run, walking unlimited;
  * 3: moderate, unable to run, limited walking without help;
  * 4: severe, walking with one stick;
  * 5: walking with two sticks;
  * 6: unable to walk, requiring wheelchair;
  * 7: confined to the bed.
  * Interpretation: Higher scores indicate worse functional status (worse outcome).
MMSE scores | 10 years
  Mini-Mental State Examination (MMSE) is a brief screening tool used to assess cognitive function, including orientation, registration, attention and calculation, recall, and language. It is widely employed to detect cognitive impairment and monitor changes in cognitive status over time in various neurological disorders.
  * Minimum value: 0
  * Maximum value: 30
  * Interpretation: Higher scores indicate better cognitive function (better outcome).
MoCA scores | 10 years
  Montreal Cognitive Assessment (MoCA) is a more sensitive tool than MMSE for detecting mild cognitive impairment. It assesses multiple cognitive domains, including attention, concentration, executive functions, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. It is particularly useful in identifying early cognitive changes in neurodegenerative diseases.
  * Minimum value: 0
  * Maximum value: 30
  * Interpretation: Higher scores indicate better cognitive function (better outcome; typically, a score ≥26 is considered normal).
Disease-associated pathogenic genomic variants | Until the patient's causative variant(s) is definitively identified.
  By utilizing human genomic DNA research techniques such as polymerase chain reaction, Sanger sequencing, next-generation sequencing, and long-read sequencing, the reasonable pathogenic variants (including tandem repeat expansions, conventional sequencing variants, and copy number variations, etc.) that cause the symptom spectrum in particpants are identified and reported, in accordance with the guidelines of the American College of Medical Genetics and Genomics (ACMG) and the Human Genome Variation Society (HGVS).
Disease-causative genes | Until the patient's causative gene(s) is definitively identified.
  The participants' causative genes harboring pathogenic variants are reported in accordance with the guidelines established by the HUGO Gene Nomenclature Committee (HGNC).
Serum neurofilament light chain levels | 10 years
  Serum neurofilament light chain levels in participants are measured using single-molecule array (Simoa) technology.
Genome-wide methylation profiles in peripheral blood leukocytes | 10 years
  Genome-wide methylation profiles of participants will be measured using whole genome bisulfite sequencing (WGBS). The analysis will quantify methylation levels across all CpG sites in the genome of peripheral blood leukocytes, with methylation level defined as the ratio of methylated cytosines to total cytosines (methylated + unmethylated) at each CpG site. Genome-wide methylation profiles will be reported as the respective or average methylation ratio across all profiled CpG sites, with data normalized according to the ENCODE Consortium guidelines for WGBS data.

CONTACTS AND LOCATIONS:
Overall Officials: Zhi-Ying Wu, M.D&Ph.D, Study Chair — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (2):
- China (2):
  - Second Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Huashan Hospital, Fudan University, Shanghai

IPD SHARING:
Plan to Share IPD: No